CLINICAL TRIAL: NCT06189677
Title: Creation of a Biobank of Biological Samples From Fertile Men
Brief Title: Creation of a Biobank of Fertile Men
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Salonia, Professor, IRCCS San Raffaele
Other Study IDs: Urimales-2016
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Fertility
Keywords: Fertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biological samples from fertile men (blood, urine, feces, seminal fluid, saliva, buccal mucosa)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation of biological characteristics of fertile men — Sampling in outpatient settings, after biopsy or after surgery and collection of biological samples in fertile subjects

SUMMARY:
Collection and conservation of human biological material from fertile subjects, i.e. men with previous parenthood (normospermic men, natural fathers).

DETAILED DESCRIPTION:
The project aims to collect biological material derived both from surgical resections of the most common urological tumors and from peripheral blood or other biological fluids such as urine or seminal fluid when available. The objective of the study is to establish a biobank of human biological material, which will allow access to samples of extreme value for the pathophysiological study of the tumor, its origin, mechanisms and markers of progression, as well as the creation of this collection it will represent an extremely valuable tool for the study of individual response to therapies.

ELIGIBILITY:
Inclusion Criteria:

* Normospermic male individuals
* Naturally fertile male individuals
* Male individuals > 18 years

Exclusion Criteria:

* Non-normospermic male individuals
* Male individuals who are not naturally fertile
* Male individuals < 18 years

Ages: 18 Years to 60 Years | Sex: Male
Age Groups: Adult
Study Population: Normospermic male individuals, naturally fertile men recruited on an outpatient and day-hospital basis.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-06-16 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Prognostic role of the biological material | Baseline
  Biological signature in fertile men predicting potential therapeutic, prognostic and diagnostic biomarkers

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - IRCCS San Raffaele Hospital, Milan

IPD SHARING:
Plan to Share IPD: No